CLINICAL TRIAL: NCT04459507
Title: Registry of Palmoplantar Pustulosis (PPP) Treatment Patterns, Disease Burden and Treatment Outcomes in Japan
Brief Title: A Registry Study of Palmoplantar Pustulosis (PPP) Treatment Patterns, Disease Burden and Treatment Outcomes in Japan
Acronym: ProPuP
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108811; CNTO1959PAP4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Palmoplantar Pustulosis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Palmoplantar pustulosis (PPP): Participants treated with a new systemic therapy for their PPP, having had an inadequate response to a prior PPP therapy either as their first systemic therapy or as a switch from, or addition to, a previous systemic therapy will be observed. Participants will be treated in accordance with routine clinical practice in Japan in the outpatient specialist care setting. The primary data source for this study will be the medical records of each participant.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be administered as a part of this study. Both retrospective and prospective data will be collected. The retrospective data will be collected through participant charts and prospective data will be collected in accordance with clinical practice at the participant's clinic visits.

SUMMARY:
The purpose of this study is to describe the treatment patterns of participants receiving systemic treatment for of palmoplantar pustulosis (PPP) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of palmoplantar pustulosis (PPP) and/or pustulotic arthro-osteitis (PAO) in accordance with local clinical practice
* Has previously been prescribed treatment for PPP/PAO
* A decision has been made by the treating physician and the participant to commence treatment with a systemic PPP/PAO therapy, having been deemed to have an inadequate response to previous therapy (New users are defined as those participants to commence treatment on baseline visit date. Existing users are defined as those who commenced treatment prior to the baseline visit since 01 November 2019.)
* Must sign a participation agreement/informed consent form allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Are receiving, or have received within the past 3 months, anti-inflammatory or analgesic systemic therapy such as oral corticosteroid, disease modifying antirheumatic drug (DMARDs), non-steroidal anti-inflammatory drugs, opioids, phosphodiesterase 4 (PDE4) inhibitor, or biologics for any other indication (for example, psoriasis, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, and asthma)
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months before the start of the study or the first data collection time point
* Participation in an investigational study
* Participation in another observational study for guselkumab (including a post marketing surveillance study)
* If the only treatment they have received for PPP has been antibiotics

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants observed in this study newly initiated/will be newly initiating a systemic therapy for their PPP/pustulotic arthro-osteitis (PAO) - either as their first systemic therapy or as a switch from, or an addition to a previous therapy, having had an inadequate response and/or intolerant to prior PPP/PAO therapy. Participants will be treated in accordance with routine clinical practice in Japan in the outpatient specialist care setting.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2025-12-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Remain on Their 'Index Systemic' Therapy | Up to 4.5 Years
  Percentage of participants who remain on their 'index systemic' therapy will be reported.
Percentage of Participants Ceasing Their 'Index Systemic' Therapy | Up to 4.5 Years
  Percentage of participants ceasing their 'index systemic' therapy will be reported.
Time to Cessation of Index Systemic Therapy From Baseline | Baseline, Up to 4.5 Years
  Time to cessation of index systemic therapy from baseline will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Receiving Each 'Index Systemic' Therapy | Baseline
  Percentage of participants receiving each 'Index Systemic' therapy will be reported.
Percentage of Participants Adding a Concurrent Systemic Treatment to their 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants adding a concurrent systemic treatment to their 'index systemic' therapy will be reported.
Percentage of Participants Ceasing a Concurrent Systemic Treatment to their 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants ceasing a concurrent systemic treatment to their 'index systemic' therapy will be reported.
Time to Addition of a Concurrent Systemic Treatment to 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Time to addition of a concurrent systemic treatment to 'index systemic' therapy will be reported.
Time to Ceasing of a Concurrent Systemic Treatment to 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Time to ceasing of a concurrent systemic treatment to 'index systemic' therapy will be reported.
Percentage of Participants Changing the Dosage of their 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants changing the dosage of their 'index systemic' therapy will be reported.
Percentage of Participants Adding a Concurrent Non-Systemic Therapy to their 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants adding a concurrent non-systemic therapy to their 'index systemic' therapy will be reported.
Percentage of Participants Ceasing a Concurrent Non-Systemic Therapy to their 'Index Systemic' Therapy | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants ceasing a concurrent non-systemic therapy to their 'index systemic' therapy will be reported.
Percentage of Participants Switching to a First Subsequent Systemic Therapy Within the Follow-up Period | Every 6 Months Up to 4.5 Years
  Percentage of participants switching to a first subsequent systemic therapy within the follow-up period will be reported.
Time to Commencement of First Subsequent Systemic Therapy From Baseline | Baseline and Every 6 Months Up to 4.5 Years
  Time to commencement of first subsequent systemic therapy from baseline will be reported.
Percentage of Participants Switching to a Second Subsequent Systemic Therapy Within the Follow-up Period | Every 6 Months Up to 4.5 Years
  Percentage of participants switching to a second subsequent systemic therapy within the follow-up period will be reported.
Time to Commencement of Second Subsequent Systemic Therapy From Baseline | Baseline and Every 6 Months Up to 4.5 Years
  Time to commencement of second subsequent systemic therapy from baseline will be reported.
Mean and Distribution of Dermatology Life Quality Index (DLQI) Scores at Baseline | Baseline
  Mean and distribution of DLQI scores at baseline will be reported. DLQI instrument consists of 10 questions covering six domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and bother with psoriasis treatment). The response options range from 0, not affected at all, to 3, very much affected. This gives an overall range of 0 to 30 where lower scores mean better quality of life.
Mean and Distribution of European Quality of Life (EuroQol) Group, 5-Dimension, 5-Level (EQ-5D-5L) Scores at Baseline | Baseline
  Mean and distribution of EQ-5D-5L scores at baseline will be reported. EQ-5D-5L is a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension. A lower score indicates worse health.
Mean and Distribution of Health Assessment Questionnaire-Disability Index (HAQ-DI) Scores at Baseline | Baseline
  Mean and distribution of HAQ-DI scores at baseline will be reported. The Disability Index of the Health Assessment Questionnaire (HAQ-DI) assesses the functional status of the participant. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area where lower scores are indicative of better functioning.
Mean and Distribution of Work Productivity and Activity Impairment: General Health (WPAI:GH) Scores at Baseline | Baseline
  Mean and distribution of WPAI:GH scores at baseline will be reported. WPAI:GH questionnaire is a validated instrument to measure impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. It consists of 6-item questionnaire looks at the effect of health problems on ability to work and perform regular activities. The WPAI yields 4 types of scores: absenteeism (work time missed), presenteeism (impairment at work / reduced on-the-job effectiveness), work productivity loss (overall work impairment / absenteeism plus presenteeism) and activity impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Percentage of Participants with a Physician's Global Assessment (PGA) Score of 1 or Less (0 or 1) | Baseline and Every 6 Months Up to 4.5 Years
  Percentage of participants with a PGA score of 1 or less (0 or 1) will be reported. The PGA is used to determine the participant's overall palmoplantar pustulosis lesions at a given time point. Overall lesions will be graded based on the scale where, 0 = clear;1 = almost clear; 2 = Mild; 3 = Moderate; 4 = Severe; 5 = Very severe.
Change From Baseline in PGA Score | Baseline and Every 6 Months Up to 4.5 Years
  Change From baseline in PGA score will be reported. The PGA is used to determine the participant's overall palmoplantar pustulosis lesions at a given time point. Overall lesions will be graded based on the scale where, 0 = clear;1 = almost clear; 2 = Mild; 3 = Moderate; 4 = Severe; 5 = Very severe.
Change from Baseline in Palmoplantar Pustulosis Area and Severity Index (PPPASI) Score | Baseline and Every 6 Months Up to 4.5 Years
  The PPPASI assesses the severity of palmoplantar pustulosis lesions and their response to therapy. In the PPPASI system, the palms and soles are divided into 4 regions: the right palm, left palm, right sole, and left sole, which account for 20 percent (%), 20%, 30%, and 30%, respectively, of the total surface area of the palms and soles. Each of these areas is assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPPASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Change From Baseline in Pain Visual Analogue Scale (Pain-VAS) Score | Baseline and Every 6 Months Up to 4.5 Years
  Change from baseline in Pain-VAS score will be reported. Pain-VAS is used to measure subjective pain status. It is a unilateral scale anchored at 0 (no pain) and 10 (worst pain imaginable).
Change in Primary Location of Pain | Baseline and Every 6 Months Up to 4.5 Years
  Change in primary location of pain will be reported.
Change From Baseline in DLQI Score | Baseline and Every 6 Months Up to 4.5 Years
  Change from baseline in DLQI score will be reported. DLQI instrument consists of 10 questions covering six domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and bother with psoriasis treatment). The response options range from 0, not affected at all, to 3, very much affected. This gives an overall range of 0 to 30 where lower scores mean better quality of life.
Change From Baseline in EQ5D-5L Index Score | Baseline and Every 6 Months Up to 4.5 Years
  Change from baseline in EQ5D-5L index score will be reported. The EQ-5D-5L is a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
Change from Baseline in HAQ-DI Index Score | Baseline and Every 6 Months Up to .4.5 Years
  Change from baseline in HAQ-DI score will be reported. The HAQ-DI assesses the functional status of the participant. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area where lower scores are indicative of better functioning.
Change from Baseline in Work Productivity and Activity Impairment questionnaire (WPAI) | Baseline and Every 6 Months Up to 4.5 Years
  Change from baseline in WPAI will be reported. WPAI questionnaire is a validated instrument to measure impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. The higher the score the greater impact on productivity.
Percentage of Participants with Adverse Events (AEs) and serious Adverse Events (SAEs) | Up to 4.5 Years
  Percentage of participants with adverse events and serious Adverse Events will be reported. An adverse event is any untoward medical occurrence in a participant administered a medicinal (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. An adverse event can be any unfavorable and unintended sign (including an abnormal finding or lack of expected pharmacological action), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (39):
- Japan (39):
  - Akita University Hospital, Akita
  - Juntendo University Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hamamatsu University Hospital, Hamamatsu
  - Kansai Medical University Hospital, Hirakata
  - Hiroshima City Asa Citizens Hospital, Hiroshima
  - Seiwakai Hiroshima Clinic, Hiroshima
  - JR Sapporo Hospital, Hokkaido
  - Kita-harima Medical Center, Hyōgo
  - Teikyo University Hospital, Itabashi Ku
  - Okayama Saiseikai General Hospital, Kita-ku
  - Chikamori Hospital, Kochi
  - Kochi Medical School Hospital, Kochi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurashiki Medical Center, Kurashiki-shi
  - Kurume University Hospital, Kurume
  - Kuwana City Medical Center, Kuwana
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Toho University Medical Center, Ohashi Hospital, Meguro-ku
  - Nagoya City University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Okayama University Hospital, Okayama
  - Oita University Hospital, Ōita
  - Kindai University Hospital, Ōsaka-sayama
  - Shiga University of Medical Science Hospital, Ōtsu
  - Hokkaido University Hospital, Sapporo
  - Sasebo Chuo Hospital, Sasebo
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Shinjuku-ku
  - Takamatsu Red Cross Hospital, Takamatsu
  - St. Luke's International Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Fujita Health University Hospital, Toyoake
  - Ehime University Hospital, Tōon
  - Yokosuka Kyosai Hospital, Yokosuka

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency